CLINICAL TRIAL: NCT01004874
Title: Avastin in Combination With Radiation and Temozolomide Followed by Avastin, Temozolomide, and Topotecan for Glioblastoma Multiformes and Gliosarcomas
Brief Title: Avastin/Radiation (XRT)/Temozolomide (Temodar) Followed by Avastin/Temodar/Topotecan for Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019960
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Malignant Glioma; Glioblastoma; Gliosarcoma
Keywords: malignant glioma; glioblastoma; gliosarcoma; Avastin; bevacizumab; Topotecan; Hycamtin; Temozolomide; Temodar; Pro00019960; Vredenburgh; Duke; Desjardins
MeSH Terms: conditions — Glioma; Glioblastoma; Gliosarcoma | interventions — Bevacizumab; Temozolomide; Radiotherapy; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab, XRT, Temozolomide, Topotecan (Experimental): Patients are treated with standard radiation therapy and daily temozolomide at 75 mg/ m2 daily for 6.5 weeks of radiation. Following completion of radiation therapy, patients have a MRI and, if there is no evidence of disease progression, patients receive 12 cycles of Avastin, temozolomide, and topotecan. Beginning a minimum of 14 days after the last radiation treatment, the Avastin is dosed at 10 mg/kg every other week; temozolomide is given at 150 mg/m2 daily the first 5 days in combination with topotecan on days 2 through 6 at 1.5 mg/ m2 for patient not taking EIAEDs and 2.0 mg/ m2 for patients taking EIAEDs on days 2-6 of each 28-day.
  Interventions: Drug: Bevacizumab; Drug: Temozolomide; Radiation: Radiation Therapy (XRT); Drug: Topotecan

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (Avastin) at 10 mg/kg every other week during standard radiation therapy (XRT). Following XRT, bevacizumab will remain at 10 mg/kg every other week.
  Other Names: Avastin
Drug: Temozolomide — Daily temozolomide at 75 mg/ m2 daily for 6.5 weeks of radiation therapy (XRT). Following XRT, temozolomide will be dosed at 150 mg/m2 daily the first 5 days of each 28-day cycle.
  Other Names: Temodar
Radiation: Radiation Therapy (XRT) — Standard radiation therapy for approximately 6.5 weeks
Drug: Topotecan — Following standard radiation therapy, patients will receive topotecan on days 2 through 6 of each 28-day cycle at a dose of 1.5 mg/m2 for patients not taking enzyme-inducing anti-epileptic drugs (EIAEDs) and 2.0 mg/m2 for patients taking EIAEDs.
  Other Names: Hycamtin

SUMMARY:
This is a phase II study of the combination of radiation therapy, temozolomide and Avastin followed by Avastin, temozolomide, and topotecan in grade IV malignant glioma patients.

DETAILED DESCRIPTION:
The primary objective of this study is to use 6-month progression-free survival to assess the efficacy of the combination of radiation therapy, temozolomide and Avastin followed by Avastin, temozolomide, and topotecan in the treatment of grade IV malignant glioma patients following surgical resection. Secondary objectives are to determine the overall survival following the combination of radiation therapy, temozolomide and Avastin followed by Avastin, temozolomide, and topotecan and to describe the toxicity of radiation therapy, temozolomide and Avastin followed by Avastin, temozolomide, and topotecan.

The study will have survival and toxicity endpoints. Patients will be treated with standard radiation therapy and daily temozolomide for 6 and a half weeks of radiation. Avastin will be administered every other week beginning a minimum of 28 days after the last major surgical procedure, open biopsy, or significant traumatic injury. Following completion of radiation therapy, patients will have a MRI and if there is no evidence of disease progression, patients will receive 12 cycles of Avastin, temozolomide, and topotecan (beginning a minimum of 14 days after the last radiation treatment). Subjects will be identified by the investigator as those patients who have newly diagnosed grade 4 malignant glioma (glioblastoma multiforme or gliosarcoma), and be within 6 weeks of the last major surgical procedure, craniotomy, open biopsy, or stereotactic biopsy.

Fifty (50) patients will initially be accrued to the study and the overall efficacy of the treatment regimen assessed. Analyses will be conducted within subgroups defined by methylation status.

Early side effects of radiation that may start during radiation include hair loss, scalp redness, inflammation of the ear canals, and fatigue. There is a small chance of long-term effects from radiation, occurring after months or years after completion. These may include worsening of mental function, hearing, vision, strength and coordination. In initial Phase I and II clinical trials, four potential Avastin-associated safety signals were identified: hypertension, proteinuria, thromboembolic events, and hemorrhage. Temozolomide has been well tolerated by both adults and children with the most common toxicity being mild myelosuppression. Other, less likely, potential toxicities include nausea and vomiting, constipation, headache, alopecia, rash, burning sensation of skin, esophagitis, pain, diarrhea, lethargy, and hepatotoxicity. With topotecan, reversible myelosuppression with leukopenia and thrombocytopenia is dose limiting. Nausea and vomiting, as well as diarrhea and alopecia, are frequent. Moderate fatigue, transient elevation of hepatic transaminase levels, stomatitis, anemia, fever, mucositis, flu-like symptoms, and rash have been reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of WHO grade IV primary malignant glioma (glioblastoma multiforme or gliosarcoma). Patients have to be within 6 weeks of the last major surgical procedure.
* Age > or = to 18 years.
* An interval of at least 2 weeks and not > 6 weeks between prior major surgical procedure and study enrollment.
* No prior radiotherapy or chemotherapy for a brain tumor
* Karnofsky > or = to 60%.
* Hemoglobin ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥ 1,500 cells/microliter, platelets ≥ 125,000 cells/microliter.
* Serum creatinine ≤ 1.5 mg/dl, serum glutamic oxaloacetic transaminase (SGOT) and bilirubin ≤ 1.5 times upper limit of normal.
* Signed informed consent approved by the Institutional Review Board
* If sexually active, patients must agree to use appropriate contraceptive measures for the duration of the study and for 6 months afterwards as stated in the informed consent.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
* Active infection requiring IV antibiotics.
* Prior treatment with radiotherapy or chemotherapy for a brain tumor, irrespective of the grade of the tumor.
* Evidence of > grade 1 central nervous system (CNS) hemorrhage on baseline MRI on CT scan.

Avastin-specific Exclusion Criteria:

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study enrollment
* History of hemoptysis (≥ ½ teaspoon of bright red blood per episode) within 1 month prior to study enrollment
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation within 6 months prior to study enrollment
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria at screening as demonstrated by either urine protein:creatinine (UPC) ratio ≥ 1.0 at screening OR urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of Avastin
* Pregnant (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-12-30 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Avastin, XRT, Temodar Followed by Avastin, Temodar, Topotecan: Avastin, XRT, Temodar followed by Avastin, Temodar, Topotecan : Standard radiation therapy and daily temozolomide at 75 mg/ m2 daily for 6.5 weeks of radiation in combination with Avastin at 10 mg/kg every other week.
  This will be followed by Avastin at 10 mg/kg every other week, temozolomide at 150 mg/m2 daily the first 5 days in combination with topotecan at 1.5 mg/m2 (patients not taking enzyme-inducing anti-epileptic drugs) or 2.0 mg/m2 (patients taking enzyme-inducing anti-epileptic drugs) on Days 2-6 of each 28-day cycle.
Period: Overall Study
Arm/Group | Avastin, XRT, Temodar Followed by Avastin, Temodar, Topotecan
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avastin, XRT, Temodar Followed by Avastin, Temodar, Topotecan
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Macdonald criteria, or to death due to any cause.
Time Frame: 6 months
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Bevacizumab, XRT, Temozolomide, Topotecan: Bevacizumab, XRT, Temozolomide followed by Bevacizumab, Temozolomide, Topotecan : Standard radiation therapy and daily temozolomide at 75 mg/ m2 daily for 6.5 weeks of radiation in combination with Bevacizumab at 10 mg/kg every other week.
  This will be followed by Bevacizumab at 10 mg/kg every other week, temozolomide at 150 mg/m2 daily the first 5 days in combination with topotecan at 1.5 mg/m2 (patients not taking enzyme-inducing anti-epileptic drugs) or 2.0 mg/m2 (patients taking enzyme-inducing anti-epileptic drugs) on Days 2-6 of each 28-day cycle.
Arm/Group | Bevacizumab, XRT, Temozolomide, Topotecan
Number analyzed (Participants) | 80
percentage of participants | 88.8 [79.5 to 94.0]

2. Secondary Outcome: One and Two Year Overall Survival
Description: Time in months from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date.
Time Frame: One year and two years
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab, XRT, Temozolomide, Topotecan
Number analyzed (Participants) | 80
percentage of participants
  One year Overall Survival | 73.8 [62.6 to 82.0]
  Two year Overall Survival | 35.6 [23.9 to 47.6]

3. Secondary Outcome: Median Overall Survival
Description: OS was defined as time in months from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 27 months
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, XRT, Temozolomide, Topotecan
Number analyzed (Participants) | 80
months | 17.2 [15.5 to 21.5]

4. Secondary Outcome: Number of Patients Experiencing a Central Nervous System (CNS) Hemorrhage or a Systemic Hemorrhage
Description: Number of times a CNS hemorrhage or systemic hemorrhage was experienced
Time Frame: 27 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Bevacizumab, XRT, Temozolomide, Topotecan
Number analyzed (Participants) | 80
participants
  Grade 2 central nervous system (CNS) hemorrhage | 1
  Grade 3 CNS hemorrhage | 0
  Grade 4 CNS hemorrhage | 2

5. Secondary Outcome: Number of Patients Experiencing a Greater Than or Equal to Grade 4 Hematologic or a Greater Than or Equal to Grade 3 Non-hematologic Toxicity
Description: Number of times a grade ≥4 hematologic or grade ≥3 non-hematologic toxicity was experienced
Time Frame: 27 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Bevacizumab, XRT, Temozolomide, Topotecan
Number analyzed (Participants) | 80
participants
  Greater than equal Gr.4 hematologic toxicites | 23
  Greater than equal Gr.3 non-hematologic toxicites | 17

6. Secondary Outcome: Median Progression-free Survival
Description: PFS was defined as time in months from the start of study treatment to the date of first progression according to Macdonald criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: 27 months
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, XRT, Temozolomide, Topotecan
Number analyzed (Participants) | 80
months | 11.1 [9.4 to 13.6]

ADVERSE EVENTS:
Time Frame: 27 months
Description: Adverse events gathered in Common Terminology Criteria for Adverse Events (CTCAE) v.3.0 and converted to v.4.0 for entry into ClinicalTrials.gov.
Arm/Group | Avastin, XRT, Temodar Followed by Avastin, Temodar, Topotecan
Serious Adverse Events (participants affected / at risk) | 17/80
Other Adverse Events (participants affected / at risk) | 33/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin, XRT, Temodar Followed by Avastin, Temodar, Topotecan (N=80)
Death NOS (General disorders) | 2
Fever (General disorders) | 2
Abdominal infection (Infections and infestations) | 1
Infections and infestations - Other, specify: Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10 (Infections and infestations) | 1
Infections and infestations - Other, specify: Septic Shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 2
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 7
White blood cell decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 3
Ischemia cerebrovascular (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 4
Confusion (Psychiatric disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin, XRT, Temodar Followed by Avastin, Temodar, Topotecan (N=80)
Neutrophil count decreased (Investigations) | 17
Platelet count decreased (Investigations) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes